CLINICAL TRIAL: NCT06248762
Title: Effectiveness of a Positive Psychology and Mindfulness Based App for Parents of Children with a Neurodevelopmental Disorder (NDD): Study Protocol of a Pragmatic Randomized Controlled Trial
Brief Title: PPI and Mindfulness App for Parents of Children with a NDD
Acronym: Adappt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Twente (Other)
Responsible Party: Principal Investigator, Kim Tonis, Principal Investigator, University of Twente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: University of Twente
Record Dates: First submitted 2024-01-25; First posted 2024-02-08 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Stress; Mental Health; Mental Well-being
Keywords: ability to adapt; Adappt
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Delayed waitlist control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention condition (Experimental): Participants will use the app for 4 weeks, daily for 10-15 minutes
  Interventions: Other: Adappt
- Waitlist control condition (Other): Participants in the control condition will start using the app 4 months after the start (baseline)
  Interventions: Other: Adappt

INTERVENTIONS:
Other: Adappt — An app to support parents of children with a NDD

SUMMARY:
An app based on positive psychology and mindfulness to support the mental well-being of parents of children with a Neurodevelopmental Disorder (NDD) was developed and will be evaluated on effectiveness.

DETAILED DESCRIPTION:
This pragmatic randomized controlled trial aims to assess the effectiveness of the Adappt app, an app developed to support the mental well-being of parents of children with a neurodevelopmental disorder (NDD), such as autism and ADHD. This app was developed since research has shown that these parents experience higher stress levels than parents of typically developing children. Furthermore, the app was developed in collaboration with parents of children with a NDD, mental health care professionals and scientists in Europe.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years
2. parent of one or more children (< 18 years) diagnosed with or suspected of a NDD
3. having access to internet
4. in possession of an e-mail address,
5. in possession of a smartphone or tablet
6. willing to use the digital intervention for a month, daily for approximately 15 minutes a day.

Exclusion Criteria:

1. presence of severe anxiety symptoms
2. presence of moderately severe to severe depressive symptoms
3. being in treatment for mental health issues (the parent self)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Ability to Adapt | Change from baseline to post intervention (1 month post baseline) and first follow up (4 months post baseline)
  Measured with the10-item Generic Sense of Ability to Adapt Scale (GSAAS). An average score will be calculated ranging from 0 to 4, with higher scores being indicative of higher perceived ability to adapt.

SECONDARY OUTCOMES:
Mental well-being | Change from baseline to post intervention (1 month post baseline) and first follow up (4 months post baseline)
  Measured with the 14-item Mental Health Continuum - Short Form (MHC-SF). Averages will be calculated for mental well-being and the subscales emotional, social and psychological well-being, ranging from 0 to 5, with higher scores being indicative for more mental (social, emotional and psychological) well-being.
Stress | Change from baseline to post intervention (1 month post baseline) and first follow up (4 months post baseline)
  Measured with the-10 item perceived stress scale (PSS). Sum scores will be calculated ranging from 0 to 40, with higher scores being indicative of larger levels of perceived stress.
Anxiety | Change from baseline to post intervention (1 month post baseline) and first follow up (4 months post baseline)
  Measured with the 7-item Hospital Anxiety and Depression Scale (HADS-A). A sum score will be calculated ranging from 0 to 21, with higher scores being indicative of larger anxiety levels.
Depressive symptoms | Change from baseline to post intervention (1 month post baseline) and first follow up (4 months post baseline)
  Measured with the 9-item Patient Health Questionnaire (PHQ-9). Sum scores will be calculated ranging from 0 to 27, with higher scores being indicative for larger depressive levels.
Parenting self-efficay and behavior of child | Change from baseline to post intervention (1 month post baseline) and first follow up (4 months post baseline)
  Measured with the 24-item Child Adjustment and Parent Efficacy Scale - Developmental Disability (CAPES-DD). A sum score will be calculated for parental self-efficacy, ranging from 16 to 160, with higher scores being indicative of larger parental self-efficacy levels. A sum score will be calculated for the child behavioral subscales: emotional problems (0-4), behavioral problems (0-30), prosocial behavior (0-24) and total problems (0-48).
Savoring the moment | Change from baseline to post intervention (1 month post baseline) and first follow up (4 months post baseline)
  Measured with the 8-item savoring the moment subscale of the Savoring Beliefs Inventory (SBI). Sum scores ranging from -24 to +24 will be calculated, with higher scores being indicative of a stronger savoring in the moment.
Self-reassuring | Change from baseline to post intervention (1 month post baseline) and first follow up (4 months post baseline)
  Measured with 5-item reassuring-self subscale of the Forms of Criticism/Self-Attacking and Self- Reassuring Scale Short Form (FSCRS-SF). Sum scores ranging from 0 to 20 will be calculated, with higher scores being indicative for a larger sense of self-reassurance.
Postive aspects of caregiving | Change from baseline to post intervention (1 month post baseline) and first follow up (4 months post baseline)
  Measured with the 9-item Positive Aspects of Caregiving (PAC). A sum score will be calculated ranging from 9 to 45, with higher scores being indicative of more positive aspects of caregiving.
Psychological flexibility | Change from baseline to post intervention (1 month post baseline) and first follow up (4 months post baseline)
  Measured with the 7-item Acceptance and Action Questionnaire-II (AAQ-II). Sum scores will be calculated, ranging from 7 to 49, with higher scores being indicative for larger levels of psychological flexibility.
Positive coping skills | Change from baseline to post intervention (1 month post baseline) and first follow up (4 months post baseline)
  Measured with the (16 items of the) subscales Acceptance, Positive refocusing, Positive reappraisal, Putting into perspective of the Cognitive Emotion Regulation Questionnaire (CERQ). Sum scores ranging from 4 to 20 will be calculated for each subscale, with higher scores being indicative of larger cognitive strategy use frequency.
Mindfulness | Change from baseline to post intervention (1 month post baseline) and first follow up (4 months post baseline)
  Measured with the 15-item Mindfulness Attention Awareness Scale (MAAS). Mean scores will be calculated ranging from 1 to 6, with higher scores being indicative of more mindfulness.

OTHER OUTCOMES:
Satisfaction with the app | Satisfaction with the app will be measured post intervention. This is 1 month post baseline for the intervention condition participants and at the second follow-up (7 months after baseline) for the control condition participants.
  Measured with the 8-item Client Satisfaction Questionnaire (CSQ-8). A sum score will be calculated ranging from 8 to 32, with higher scores being indicative of a larger satisfaction with the Adappt app.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Twente, Enschede, Netherlands

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared

REFERENCES:
- [Derived] Tonis KJM, Drossaert CHC, Ten Klooster PM, Schaer M, Bourgeron T, Buitelaar JK, Sadaka Y, Freitag CM, Lapidus KM, Chiocchetti AG, Staal WG, Bohlmeijer ET. Effectiveness of a positive psychology and mindfulness-based app on mental health for parents of children with a neurodevelopmental disorder: study protocol of a pragmatic international randomized controlled trial. Trials. 2024 Jun 26;25(1):412. doi: 10.1186/s13063-024-08256-w. PMID 38926739